CLINICAL TRIAL: NCT03583528
Title: Evaluation of the Safety and Sensitivity of 68Ga-DOTATOC PET/CT for Imaging NET Patients
Brief Title: DOTATOC PET/CT for Imaging NET Patients
Status: Active, not recruiting | Type: Observational
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Other Study IDs: H17-00909
Record Dates: First submitted 2018-06-08; First posted 2018-07-11 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Neuroendocrine Tumors; Insulinoma; Gastrinoma; Glucagonoma; Vipoma; Pheochromocytoma; Paraganglioma; Neuroblastoma; Ganglioneuroma; Medullary Carcinoma; Pituitary Adenoma; Medulloblastoma; Merkel Cell Carcinoma; Small-cell Lung Cancer; Meningioma; Carcinoid
MeSH Terms: conditions — Neuroendocrine Tumors; Insulinoma; Gastrinoma; Glucagonoma; Vipoma; Pheochromocytoma; Paraganglioma; Neuroblastoma; Ganglioneuroma; Carcinoma, Medullary; Pituitary Neoplasms; Medulloblastoma; Carcinoma, Merkel Cell; Small Cell Lung Carcinoma; Meningioma; Carcinoid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PET/CT Diagnostic Imaging: Each subject will have two PET/CT scans, one using 68Ga-DOTATOC and the other using 18F-FDG. The 68Ga-DOTATOC radioactive tracer is manufactured for this study under a Clinical Trial Application filed with Health Canada. 18F-FDG is considered standard care and has been approved by Health Canada.
  Interventions: Diagnostic Test: 68Ga-DOTATOC PET/CT; Diagnostic Test: 18F-FDG PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-DOTATOC PET/CT — Blood pressure, heart rate, and oxygen saturation levels will be recorded prior to the injection and at 5 - 15 minutes after injection.
  Each study subject will have an intravenous catheter inserted. The subject will receive a bolus intravenous dose of the radiotracer from an approved study supplier site.
  The subject will rest in a comfortable chair for 60 minutes. After this uptake phase, the blood pressure, heart rate, and oxygen saturation levels will be recorded again. The subjects will then be taken to a designated washroom and asked to void prior to being scanned in order to clear excreted radiotracer activity from the urinary tract.
  Subjects are positioned supine, arms down, and centered on the scanner bed and the PET/CT images will be acquired.
Diagnostic Test: 18F-FDG PET/CT — 18F-FDG PET/CT For 18F-FDG as fasting period of 6 hours is required before the scan.
  Each study subject will have an intravenous catheter inserted. The subject will receive a bolus intravenous dose of the radiotracer from an approved study supplier site.
  The subject will rest in a comfortable chair for 60 minutes. The subjects will then be taken to a designated washroom and asked to void prior to being scanned in order to clear excreted radiotracer activity from the urinary tract.
  Subjects are positioned supine, arms down, and centered on the scanner bed and the PET/CT images will be acquired.

SUMMARY:
Neuroendocrine tumours (NETs) are generally slow growing, but some can be aggressive and resistant to treatment. Compared to healthy cells, the surface of these tumor cells has a greater number of special molecules called somatostatin receptors (SSTR). Somatostatin receptor scintigraphy and conventional imaging are used to detect NETs.

This study proposes 68Gallium(68Ga)-DOTATOC positron emission tomography/computed tomography (PET/CT) is superior to current imaging techniques. The goal is to evaluate the safety and sensitivity of 68Ga-DOTATOC PET/CT at detecting NETs and other tumors with over-expression of somatostatin receptors.

DETAILED DESCRIPTION:
Each subject will have two PET/CT scans, one using 68Ga-DOTATOC and the other using 18-Fluoride-Fluorodeoxyglucose (18F-FDG). The 68Ga-DOTATOC radioactive tracer is manufactured for this study under a Clinical Trial Application filed with Health Canada. 18F-FDG is considered standard care and has been approved by Health Canada.

After providing informed written consent subjects will complete a medical history questionnaire.

Monitoring of adverse events There will be short-term evaluation of adverse events by comparison of vital signs before and after administration of 68Ga-DOTATOC. Twenty-four hours after 68Ga-DOTATOC administration the study coordinator will call the patient and see if they have experienced any adverse events during that time period and complete the adverse event questionnaire found in section 9.6.

Follow-up Assessments

The following information will be collected up to 3 years following the PET/CT scans:

* Initiation of a new treatment
* Laboratory results and pathology reports
* Results of imaging studies
* Final clinical diagnosis by physician and relevant clinical notes

The study is expected to take approximately 4 years for accrual.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* World health organization performance status 0-2
* Able to provide written informed consent/assent (or consent by guardian for subjects <19 years)
* Patients must be able to tolerate the physical/logistical requirements of completing a PET scan including lying flat for up to 30 minutes and tolerating intravenous cannulation for injection.

Patients must require imaging for either staging or re-staging of:

* Gastroenteropancreatic tumors (e.g. carcinoids, gastrinoma, insulinoma, glucagonoma, VIPoma, etc.), functioning and non-functioning
* Sympathoadrenal system tumors (phaeochromocytoma, paraganglioma, neuroblastoma, ganglioneuroma)
* Medullary thyroid carcinoma
* Pituitary adenoma
* Medulloblastoma
* Merkel cell carcinoma
* Small-cell lung cancer (mainly primary tumors)
* Meningioma
* Or any other NET / with potential for overexpression of SSTR

Exclusion Criteria:

* Pregnancy
* Patients who are medically unstable ex: acute cardiac or respiratory distress, hypotensive
* Patients who exceed the safe weight limit of the PET/CT bed (204.5 kg) or who cannot fit through the PET/CT bore (diameter 70cm).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a prospective, open-label trial in patients with suspected or proven SSTR positive tumors.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-07-11 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of 68Ga-DOTATOC PET/CT in the diagnosis of SSTR positive tumors. | 3 years
  Determination of sensitivity of both exams when compared with pathology reports (if available) and compared with routine imaging (CT, MRI, Octreoscan™, US) if available and will be determined by confidence intervals using an exact binominal distribution by comparing the 68Ga-DOTATOC PET/CT with 18F-FDG and conventional imaging (if available).
  The gold standard for the detection of lesions will be established through a combination of: 1) pathology; 2) unequivocal correlative imaging results as assessed independently by 2 physicians; 3) disease progression of specific findings upon follow-up, up to three years from baseline examination; 4) a clearly unequivocal plurimetastatic pattern confirmed by any imaging modality at any of the involved sites; 5) response of lesions on subsequent imaging following therapy.

SECONDARY OUTCOMES:
Number of participants with 68Ga-DOTATOC-related adverse events as assessed by abnormal vital sign measurement. | 1 hour
  Vital signs (blood pressure, heart rate and pulse oximetry) will be measured at three time points (before and after injection, and 1 hour after the injection). All values that fall outside of the normal parameters will be assessed by a physician and reported as an adverse event.
Number of participants with self-reported 68Ga-DOTATOC-related adverse event | 24 hours
  Patients will be contacted by phone 24 hours after the 68Ga-DOTATOC PET/CT scan to see if they experienced any adverse events. These are recorded and evaluated for severity and likelihood they are related to the study drug. All adverse events will be recorded and summarized in the final report.
Total number of lesions per anatomic location identified by 68Ga-DOTATOC PET/CT | 3 years
  All lesions will be tabulated and classified by compartment (pancreas, liver, bowel, lung and mediastinum, abdomen and retroperitoneal lymph nodes, bone, other) for all imaging modalities that have been done for that subject. A total number of lesions (for all modalities) will be calculated and a proportion of lesions detected by each modality will be reported and will be compared by calculating the median and its confidence interval. This will assess the efficacy of 68Ga-DOTATOC PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Benard, MD, Principal Investigator — BC Cancer
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No